CLINICAL TRIAL: NCT07189104
Title: SAGA for Toddlers. Supporting Children's Linguistic and Socio-Emotional Development in Early Childhood Education and Care
Acronym: SAGA-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Swedish Cultural Foundation in Finland (Unknown)
Responsible Party: Principal Investigator, Mirjam Kalland, Professor, University of Helsinki
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 58/2025
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Social Emotional Competence; Language Development
Keywords: social-emotional development; language development; intervention; toddlers; early childhood education and care; caregivers; mentalization theory; SAGA model; group intervention; shared reading intervention

STUDY DESIGN:
Intervention Model Description: This is a wait-list controlled cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAGA for Toddlers intervention (Experimental): The SAGA for Toddlers intervention.
  Interventions: Behavioral: SAGA for Toddlers
- Control group (No Intervention): The personnel of the waitlist control-group will receive the intervention training after the data-collection is finished.

INTERVENTIONS:
Behavioral: SAGA for Toddlers — SAGA for Toddlers includes training sessions and workshops for the ECEC personnel on the mentalization-based shared reading intervention following the SAGA model. During the intervention shared reading sessions (5-10-minutes each) are held for groups of 2 to 3 children for 10 weeks (at least 3 sessions per week) at the ECEC by the personnel. Caregivers are involved in the intervention via caregiver meetings held at the ECEC by the investigators.
  Arms: SAGA for Toddlers intervention

SUMMARY:
The goal of this study is to investigate whether a shared reading intervention including emotion and mind-related dialogues (SAGA for Toddlers) supports the development of 11 to 36 moth-old-children in early childhood education and care.

The main questions it aims to answer are:

1. Does the SAGA model support children's social-emotional development?
2. Does the SAGA model support children's language development?

The participating children will attend the intervention at the early childhood education and care.

The participating personnel at the early childhood education and care will receive training, implement the intervention, and answer questionnaires.

The participating caregivers will attend caregiver-evenings and answers questionnaires.

DETAILED DESCRIPTION:
Background:

The SAGA intervention model is based on mentalization theory, and it aims at supporting children's social-emotional development. The intervention includes regular shared reading sessions (at least three times a week) with children in small groups held by early childhood education and care (ECEC) professionals. The personnel receive training on the method and support on organizing the reading sessions. The SAGA model has been found to support children's prosocial behavior and reduce externalizing and internalizing problems. The research has also showed a connection between children's social-emotional and language development.

The first thousand days of a child's life are the most important for their development. In early childhood education and care, the integration of care and learning, places particularly high demands on educational quality and the pedagogues' competence to support children's emotional security, language, conceptual development, and exploratory learning as an organic whole. SAGA for Toddlers aims to use the SAGA model to strengthen the identification and naming of emotions in small groups of 11 to 36-month-old children. Stories in picture books meant for very young children that touch on emotions are selected for the sessions, and mentalization-based dialogue cards and emotion cards are used for the stories to support the discussions.

SAGA for Toddlers emphasizes the importance of relationship skills and to support caregivers' understanding of the importance of early years and shared reading of picture books with their children. This is achieved not by demanding parents to provide "more" for their children, which can increase parental stress, but by supporting parents in offering a daily routine with calmer presence, free-flowing time, shared moments and reading aloud. The SAGA for Toddlers intervention also includes caregivers´ evenings held at the ECEC premises with a simple meal plus a SAGA session to strengthen co-operation with caregivers in an easily accessible way.

Aims:

The main aim of this randomized controlled trial is to investigate whether the SAGA for Toddlers model is effective in supporting 11 to 36-month-old children's 1) social-emotional and 2) language development at Swedish speaking ECEC in Finland.

In addition, the study focuses on:

3) Does the SAGA for Toddlers intervention support ECEC personnel's mentalizing abilities? 4) Does the SAGA for Toddlers intervention support caregiver's mentalizing abilities and emotional availability? 5) Does the SAGA for Toddlers intervention impact children's screen time? 5) What factors related to the child, caregivers and the ECEC personnel mediate or moderate the effectiveness of the SAGA for Toddlers intervention?

Participants and training:

ECEC centers are invited to participate in the study aiming to recruit 120 11 to 36-month-old children and their caregivers. From these centers half are randomized to receive the SAGA for Toddlers intervention and half are randomized to a waitlist control group.

The personnel of the intervention group will receive training to carry out the intervention at the ECEC, the waitlist control group will receive the intervention training after the data collection is finished. The intervention period will last for 10 weeks, including at least three SAGA for Toddlers intervention sessions per week.

The ECEC groups are offered support in the form of a resource teacher (master student/PhD student) who supports the centers in using the SAGA model and integrating it into their activities. Parents' evenings are held once before the intervention (an information session online or at the ECEC) and twice during the intervention (a workshop at the ECEC premises).

Data collection:

Data is collected 1) before the intervention, 2) during the 10-week intervention, 3) immediately after the intervention, and 3) in 1-year follow-up (1 year after the baseline measurement).

In addition to the outcome measures, the child's and caregivers' background is enquired with a background questionnaire before the intervention, including child age and gender, caregiver education, subjective economic situation, family structure, number of siblings, siblings' age, child's language skills and languages spoken at home, child's ECEC start age, age when child started to speak in sentences, screen time, hobbies and their frequency and start time, and amount of time spent reading aloud together.

Personnel's background is also enquired before the intervention, including gender, age, working experience, job title, current work tasks, education, and subjective economic situation.

ELIGIBILITY:
Inclusion Criteria:

* 11 to 36 -months old at the start of the study
* Living in Finland
* Attending Swedish speaking early childhood education and care

Exclusion Criteria:

* None

Ages: 11 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Social Emotional development | 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) In 1-year follow-up
  Social Emotional development is assessed by the personnel and caregivers with the 42-item Brief Infant-Toddler Social Emotional Assessment (BITSEA). The assessment includes two subscales Problem scores (31 items, range 0-62, higher scores indicate more problems) and Competence scores (11 items, range 0-22, higher scores indicate better social-emotional competence).
Language development | 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) In 1-year follow-up
  Language development is reported by the caregivers using the MacArthur-Bates Communicative Development Inventory (MCDI), with separate questionnaires for 8- to 16-month-old, 16- to 30 month-old, and 2,5 to 4 year-old children, correct questionnaire is chosen based on the child's age. The questionnaires measure the size of the child's expressive vocabulary, and the child's use of gestures, sentences and grammar.
Pro-social behavior | Before the intervention, 2) Immediately after the 10-week intervention, 3) In 1-year follow-up
  Pro-social behavior is assessed by the personnel and the caregivers with the 10-item child prosocial behavior questionnaire (CPBQ). The questionnaire including three subscales Comforting (range 1-15), Sharing (range 1-20), and Helping (range 0-15), higher scores indicate positive outcome.

SECONDARY OUTCOMES:
Caregiver's emotional availability | 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) In 1-year follow-up
  Caregiver's emotional availability is measured with the 36-item Emotional Availability Self-Report (EA-SR). Following Salo and colleagues (2025) three subscales are calculated: Caregiver scale (12-items, range 8 to 60), Child scale (9-items, range 9 to 45), and Dyadic scale (15-items, range 15 to 75). Higher scores indicate better outcome.
Personnel mind-mindedness | 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) In 1-year follow-up
  Personnel mind-mindedness is an index of mentalization ability. It is assessed with the mind-mindedness task. In this task, the pedagogue randomly selects four children from the children participating in the study, and freely describes them. The descriptions are audio-recorded and later transcribed. Each description will be analyzed using the coding system, which categorizes all the comments in the following categories: physical; behavioral; mental; self-referential; relational; general. A score will be obtained by calculating the number of attributes in each category. A total score (MM_TOT) will also be computed. It is assumed that more mental descriptions will indicate better mind-mindedness.
Caregiver's mentalizing ability | 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) In 1-year follow-up
  Caregiver mentalizing is self-assessed with the 24-item Parental Mentalizing Questionnaire. The measure has four subscales: 1) Parental self-mentalizing ("SELF", 7 items, range: 7-49), 2) Parental child-mentalizing ("CHILD", 7 items, range: 7-49), 3) Lack of Effort ("LE", 5 items, range: 5-35), and 4) Curiosity ("C", 5 items, range: 5-35). Higher scores on the SELF, CHILD, and C subscales, and a lower score on the LE subscale indicate better outcome.
Personnels' mentalizing ability | 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) In 1-year follow-up
  Personnels' mentalizing ability is self-assessed with the 28-item Mentalization Scale (MentS). MentS has three subscales: MentS-Self (MentS-S, 8 items, range 1-40) and MentS-Others (MentS-O, 10 items, range 10-50) assessing the ability to mentalize one self's or other people's minds, and MentS-Motivation (MentS-M, 10 items, range 10-50) assessing the respondent's motivation to mentalize about other people. Higher score means better outcome.
Child's screen time | 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) At 1-year follow up
  Child's screen time (hours per week) in 1) playing games, 2) watching content directed to children, 3) watching content directed to adults, and 4) other screen time, are enquired with a tailored questionnaire. Total screen time is calculated by summing the four types of screen time.
Application names (screen time) | Time Frame: 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) At 1-year follow up
  Application names used for video screen time and playing games with digital devices are enquired with a tailored questionnaire.
Screen time language | Time Frame: 1) Before the intervention, 2) Immediately after the 10-week intervention, 3) At 1-year follow up
  Language primarily used for video screen time and playing games with digital devices are enquired with a tailored questionnaire.

OTHER OUTCOMES:
Content of the reading sessions | After each session, during the intervention (10 weeks)
  Content of the reading sessions are enquired after each session with a session log (which book was used, did the child interact with the material). Session logs are filled by the intervention group personnel regarding the intervention sessions and by the control group personnel regarding 'business-as-usual' shared reading sessions at the group.
Number of sessions participated | After each session during the intervention (10 weeks)
  The session log is used to record the number of shared reading sessions participated by each child during the intervention
Fidelity to the intervention | During the intervention at week 1, week 5, and week 10.
  Fidelity to the SAGA for toddlers intervention model will be assessed via video recordings. The videos are analyzed qualitatively to assess how well the personnel follow the SAGA model in their interaction.
Use of the SAGA model after the active intervention at ECEC | At 1-year follow-up
  Personnel's use of the SAGA model after the 10-weeks intervention period is enquired with a questionnaire detailing the average frequency and duration of the sessions.
Use of the SAGA model at home | 1) Immediately after the 10-week intervention, 2) At 1-year follow-up
  Caregivers' use of the SAGA model in shared reading sessions with their children is enquired with a questionnaire detailing the average frequency and duration of the sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Helsinki, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Citation: Kalland, M., Linnavalli, T., & von Koskull, M. (2022). SAGA-supporting social-emotional development in early childhood education. The development of a mentalizing-based intervention. Education Sciences, 12(6), Article 409. https://doi.org/10.3390/educsci12060409
- [Background] Citation: Kalland, M., & Linnavalli, T. (2023). Associations between social-emotional and language development in preschool children. Results from a study testing the rationale for an intervention. Scandinavian Journal of Educational Research, 67(5), 791-804. https://doi.org/10.1080/00313831.2022.207092
- [Background] Martikainen, S., Kalland, M., Linnavalli, T., Kostilainen, K., Aittokoski, M., Reunamo, J., … Tervaniemi, M. (2024). Supporting social-emotional development in early childhood education and care - a randomized parallel group trial evaluating the impact of two different interventions. Scandinavian Journal of Educational Research, 68(5), 1069-1087. https://doi.org/10.1080/00313831.2023.2204119
- [Background] Linnavalli, T., Martikainen, S., Belfrage, F., & Kalland, M. (2024). SAGA: results of a second trial testing a mentalizing-based reading intervention on children and staff in early childhood education. Frontiers in Education, 9. https://doi.org/10.3389/feduc.2024.1284474